CLINICAL TRIAL: NCT05259449
Title: Efficacy of a Nutritional Education Strategy and Role of Physical Exercise on the Regulation of Appetite and Body Composition Through the Profile of Exosomes in Type 2 Diabetics (The APETEX Project)
Brief Title: Efficacy of Educational Nutrition and Exercise on the Regulation of Appetite Through Exosomes in Type 2 Diabetics
Acronym: APETEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The APETEX project; PID2020-120034RA-I00/AEI/10.13 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2021-12-17; First posted 2022-02-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin Sensitivity; Appetite regulation; aerobic exercise; Extracellular vesicles
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The project is a randomized controlled clinical trial in individuals with T2DM and obesity
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ND-INACT (No Intervention): Participants who do not receive either nutritional intervention or an exercise program. They will be instructed to maintain their normal life habits with respect to physical activity and diet.
- Moderate-intensity continuous training (ND-MICT) (Active Comparator): Participants who do not receive nutritional intervention but are enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Other: Moderate-intensity continuous training (MICT)
- High-intensity interval training (ND-HIIT) (Active Comparator): Participants who do not receive nutritional intervention but are enrolled in a high-intensity interval training exercise program.
  Interventions: Other: High-intensity interval training (HIIT)
- Nutritional Intervention (D-INACT) (Active Comparator): Participants who receive nutritional intervention but not an exercise program.
  Interventions: Behavioral: Nutritional Intervention
- Nutritional Intervention Moderate-intensity continuous training (D-MICT) (Experimental): Participants who receive nutritional intervention and are enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Behavioral: Nutritional Intervention; Other: Moderate-intensity continuous training (MICT)
- Nutritional Intervention High-intensity interval training (D-HIIT) (Experimental): Participants who receive nutritional intervention and are enrolled in a high-intensity interval training exercise program.
  Interventions: Behavioral: Nutritional Intervention; Other: High-intensity interval training (HIIT)

INTERVENTIONS:
Behavioral: Nutritional Intervention — The nutritional intervention was conducted through biweekly (± 3 days) in-person consultations with a nutritionist or dietitian. Firstly, the patient's diet was analyzed. Then, participants were guided to follow a Mediterranean pattern-based and mildly calorie-restricted diet, with the primary goal of achieving a 5 % reduction in body weight and reducing blood glucose levels. Meal plans were created using Nutrium® software , personalized to each participant's lifestyle and food preferences, and reviewed at each biweekly consultation. The dietary plan included at least 4 meals per day, ensuring a well-distributed intake of carbohydrates, a balanced distribution of macro- and micronutrients, and the inclusion of foods rich in prebiotics and probiotics. Moreover, some suggestions about the combination of foods and culinary techniques were provided. Only one session through the intervention was allowed to be attended telephonically.
  Arms: Nutritional Intervention (D-INACT); Nutritional Intervention High-intensity interval training (D-HIIT); Nutritional Intervention Moderate-intensity continuous training (D-MICT)
Other: High-intensity interval training (HIIT) — Participants assigned to the HIIT completed 3 weekly sessions, with 1-2 days of rest between sessions, on a cycle ergometer for 12 weeks. The training load (TL) was determined from an incremental test until volitional exhaustion with one-minute work intervals (from 85% to 165% of maximal power output during VO2max test [Wmax] and with 10% increments) separated by 1.5-minute rest periods (at 20% Wmax). The program consisted of a 3 minutes warm-up with the first 2 minutes at 20% and last minute at 40% of the TL, followed by 10 series of 1 min duration at 90% of TL, with 1 minute of rest between sets at 20% of TL and ending with 2 minutes of cool-down at 20% of TL (estimated total time of the session: 25 minutes). A 5% increase in workload was applied when, for two consecutive sessions, the first three intervals failed to exceed 85%, and the last five did not reach 90% of maximal HR. Participants were asked to maintain a cadence above 80RPM.
  Arms: High-intensity interval training (ND-HIIT); Nutritional Intervention High-intensity interval training (D-HIIT)
Other: Moderate-intensity continuous training (MICT) — Participants assigned to the MICT completed 3 weekly sessions, with 1-2 days of rest between sessions, on a cycle ergometer for 12 weeks. The MICT program consisted of 50 minutes of continuous pedaling at an intensity approximately 10 % above the lactate threshold, with cadence maintained between 60-80 rpm. The training load was increased by 10% if these two conditions were met: 1) no increase of at least 2 beats of heart rate from minute 20 to minute 40 of the training session, and 2) lactate levels below 2 mmol/L in minute 48 of the session. The training load for the first session was determined by an adjustment test consisting of an incremental test with five consecutive 10-minute phases at a constant cadence (60-80 RPM) from 90% to 130% of the ventilatory threshold power, calculated from the FatOx test data, with 10% increments in each step. was determined by the phase in which HR increased by ≥ 3 beats between phases and blood lactate levels increased by ≥ 1 mmol/L between phases.
  Arms: Moderate-intensity continuous training (ND-MICT); Nutritional Intervention Moderate-intensity continuous training (D-MICT)

SUMMARY:
The aim of this randomized controlled trial is to investigate the effects of different aerobic modalities; moderate-intensity continuous training (MICT) and high-intensity interval training (HIIT), and a nutritional intervention (D) on appetite regulation, appetite-related hormones, neural responses to food cues (EEG), and exosome-derived molecular signals in patients with type 2 diabetes (T2D) and obesity. It will also examine whether these effects differ between men and women.

The main questions it aims to answer are:

* What is the isolated and combined effect of these exercise modalities and diet on glucose metabolism, insulin dynamics, miRNA exosomal expression, appetite hormones, and neural responses to food stimuli?
* Is there a sex-specific best combination choice for improving appetite regulation and metabolic control?
* Are changes in miRNA exosomal profile, appetite-related hormones, and EEG-based neural responses associated with other health-related outcomes such as body composition, fat mass reduction, insulin sensitivity, physical condition, and quality of life?

To answer these questions, researchers designed a two-factor study. One factor was diet, with two levels Diet (D) and no diet (ND). The second factor was exercise, with three levels (inactive (INACT), MICT, and HIIT). Participants were randomly allocated into six groups: ND-INACT, ND-MICT, ND-HIIT, D-INACT, D-MICT, and D-HIIT.

Participants will:

* Undergo a 12-week intervention within their assigned group.
* Visit the research facilities three times per week if assigned to an exercise group, or once every two weeks if in a diet group.

DETAILED DESCRIPTION:
This randomized controlled trial is conducted in the Province of Cádiz (Spain). A total of 146 participants with type 2 diabetes (T2D) and obesity were enrolled and underwent baseline and post-intervention assessments of the study outcomes. Immediately after baseline evaluations, participants were randomly allocated to one of the six study groups. Randomization was stratified by sex to ensure approximately 50% of participants in each group were women. All participants received detailed written and verbal information about the study objectives, procedures, benefits, and potential risks before providing written informed consent. The study complied with the Declaration of Helsinki and was approved by the Research Ethics Committee of Cádiz (registration number 92.21; PEIBA number 1026-N-21) and by the Coordinating Committee for Biomedical Research Ethics of Andalusia (registration number 92.21; PEIBA number 1026-N-21; internal codes SICEIA-2025-001870 and SICEIA-2025-000778).

At both baseline and post-intervention, participants attended the research facilities in the morning following an overnight fast and were instructed to maintain their usual lifestyle while avoiding alcohol, caffeine, and strenuous physical activity for the specified periods prior to testing. During these visits, a comprehensive set of assessments was conducted to capture the effects of the interventions across multiple domains. These included measures of glucose metabolism, insulin dynamics, plasma exosomal miRNA expression, appetite-regulating hormones, neural responses to food cues, subjective appetite, body composition, dietary intake and adherence, physical activity and sedentary behavior, resting and maximal fat oxidation, cardiorespiratory fitness, blood pressure, and self-reported quality of life. Post-intervention assessments followed the same protocol, with participants in exercise groups completing their final training session at least 72 hours before testing. This design allows evaluation of both the isolated and combined effects of exercise and diet interventions on physiological, molecular, behavioral, and lifestyle outcomes, as well as potential sex-specific differences in response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D or prediabetes (HbA1c ≥ 5.7%)
* No history of substance abuse (tobacco, alcohol, or other drugs).
* Body mass index >25 kg/m², maintaining the habitual dietary patterns with stable body weight for at the least 6 months
* Stable physical activity and medication regimen for at least 6 months
* Not insulin-dependent
* Absence of injury, disease, disability, or other known medical condition which could affect the ability to successfully participate in physical exercise tests
* Absence of tumours and cancer disease
* Absence of other pathologies that could affect the study outcomes.
* Not under medication regimen that could affect the study outcomes.
* Being able to understand a communication in Spanish or English.
* Not pregnant

Exclusion Criteria:

* Failure to attend more than 2 consecutive or a total of 4 sessions of nutritional intervention.
* Failure to attend more than 4 consecutive or a total of 6 sessions of physical training.
* Serious injury
* Voluntary withdrawal
* Increased dose of diabetes medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Assessed changes in Glucose concentration | Pre and Post the 12-week intervention
  Glucose concentration (mg/dL) was measured from blood samples collected from the antecubital vein after at least 8 hours of fasting and at 30, 60, 90, 120, and 180 minutes after the ingestion of 75 grams of glucose (Nuter-tec, 75 g/200 mL, orange flavor). Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine consumption for 24 hours, and avoid vigorous physical activity for 72 hours. Blood samples were centrifuged at 4000 rpm for 7 minutes, and serum was analyzed. Glucose concentrations were determined using the colorimetric method performed on the Alinity CI system (Abbott Laboratories, Abbott Park, IL, USA).
Assessed changes in Insulin concentration | Pre and Post the 12-week intervention
  Insulin concentration (µU/mL) was measured from blood samples collected from the antecubital vein into serum separator tubes after at least 8 hours of fasting and at 30, 60, 90, 120, and 180 minutes after the ingestion of 75 grams of glucose (Nuter-tec, 75 g/200 mL, orange flavor). Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine consumption for 24 hours, and avoid vigorous physical activity for 72 hours. Blood samples were centrifuged at 4000 rpm for 7 minutes, and serum was analyzed. Insulin concentrations were determined by chemiluminescent immunoassays performed on the Alinity CI system (Abbott Laboratories, Abbott Park, IL, USA).
Assessed changes in Insulin Resistance: HOMA-IR | Pre and Post 12-week intervention
  Insulin resistance was estimated using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), calculated as fasting insulin (µU/mL) multiplied by fasting glucose (mg/dL) divided by 405.
Assessed changes in Insulin Sensitivity: Matsuda Index | Pre and Post 12-week intervention
  Whole body insulin sensitivity was estimated through the Matsuda Index, calculated as 10,000 / √[(fasting glucose (mg/dL) × fasting insulin (µU/mL)) × (mean glucose during Oral Glucose Tolerance Test (mg/dL) × mean insulin during Oral Glucose Tolerance Test (µU/mL))].
Assessed changes in Insulin Sensitivity: Quicki | Pre and Post 12-week intervention
  Insulin sensitivity was estimated through the Quantitative Insulin Sensitivity Check Index (QUICKI), calculated as 1 / [log(fasting insulin (µU/mL)) + log(fasting glucose (mg/dL))].
Assessed changes in Plasma Exosomal miRNA expression | Pre and Post the 12-week intervention
  Fasting blood samples (fast 8-10 hours) were centrifuged (1500×g, 15 min, 4 °C) and the resulting plasma was divided into aliquots (500 µL) and stored at -80°C. Exosomes will be isolated from 600 µL of plasma using the miRCURY Exosome Kits (Qiagen, Netherlands). Total RNA was extracted from 200 μL of exosome samples using the miRNeasy Serum/Plasma Advanced Kit (Qiagen). Reverse transcription was performed with the miRCURY LNA RT Kit, incubated at 42°C for 60 min, 95°C for 5 min, and stored at -20°C. Quantitative PCR was carried out using the miRCURY LNA SYBR Green PCR Kit and miRNA-specific assays on a CFX Connect System (Bio-Rad). MiRNA expressions (Cq values) were normalized using reference miRNAs. Relative expression was determined with the 2^-ΔCq method, and fold changes were calculated using the 2^-ΔΔCq method, ensuring accurate quantification of miRNA expressions from exosomal RNA.
Assessed changes in Appetite hormones | Pre and Post the 12-week intervention
  Appetite-regulating hormones will be assessed from blood samples collected after an 8-10-hour overnight fast, with participants seated at rest for 15 minutes. Fasting samples will be drawn from the antecubital vein using EDTA tubes for appetite hormones and CAT tubes for serum cortisol. EDTA tubes will be inverted, centrifuged at 1500 × g for 15 minutes at 4 °C, and plasma aliquoted into 500 µL tubes with 5 µL protease inhibitors, then stored at -80 °C. Ghrelin, leptin, GLP-1, and GIP will be measured fasting and 90 minutes post-75 g glucose using the MILLIPLEX® Metabolic Hormone Panel V3 with a Luminex® xMap system; intra- and inter-assay CVs <10% and <20%. Cortisol from CAT tubes allowed to clot 30 minutes, centrifuged at 2000 × g for 10 minutes at 4 °C, aliquoted into 200 µL tubes, stored at -80 °C, and quantified using one-step CMIA on Alinity CI; emitted light inversely reflects cortisol, range 1-59.8 µg/dL, intra- and inter-assay variation <10%.
Assessed changes in task of emotional reactivity to food images | Pre and Post the 12-week intervention
  Emotional reactivity to food images will be measured using a high-density 128-channel EEG system (HydroCel Sensor Net, EGI, Inc.) during both resting state and a visual-attentional cognitive task. EEG caps will be fitted according to standardized landmarks (GND at the forehead, REF at the vertex, lateral electrodes at the eyebrows and top of ears, posterior electrode at the occipital bone), with impedance checked and adjusted by pipetting or gentle repositioning. Participants will be seated 60-70 cm from a 15'' monitor in dim lighting, with eyes aligned to the center of the screen. A 4-minute eyes-open resting-state recording will be conducted to assess baseline alpha activity (8-14 Hz). The experimental task will present images in blocks with breaks, including high- and low-calorie foods, non-food controls, and, in a separate task, images categorized as beneficial or harmful for gut microbiota based on fiber, prebiotic/probiotic content, caloric density, fat, and meat content.
Assessed changes in Appetite assessment. | Pre and Post the 12-week intervention
  Since appetite feelings modulate nutritional behavior, evaluating appetite among the intervention groups can improve the study's quality from a comprehensive perspective. After an 8-10 hour fasting period, a Visual Analogue Scale (VAS) will be completed to measure the participant's morning appetite. Likewise, they will be evaluated 90 minutes into the Oral Glucose Tolerance Test (OGTT) and at the end of it. The VAS is a valid measurement instrument for assessing the feeling of appetite.
Assessed changes in Body Weight | Pre and Post the 12-week intervention
  Body weight (kilograms, kg) was measured using a multifrequency bioelectrical impedance device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed in Height | Pre and Post 12-week Intervention
  Height (meters, m) was measured using a wall-mounted stadiometer (TANITA-LEICESTER HR-001, Tanita Corp., Tokyo, Japan) with participants standing in accordance with the manufacturer's instructions.
Assessed changes in Body Mass Index | Pre and Post 12-week Intervention
  Body Mass Index (BMI) in kilograms per square meter (kg/m²) was calculated as body weight (kg) divided by height squared (m²).
Assessed changes in Fat Mass (kilograms of Fat Mass) | Pre and Post 12-week Intervention
  Fat mass (kilograms, kg) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat Mass (percentage of Fat Mass) | Pre and Post 12-week Intervention
  Fat mass (percentage of total body weight, %) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat-free Mass (kilograms of Fat-free Mass) | Pre and Post 12-week Intervention
  Fat-free mass (kilograms, kg) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Fat-free Mass (percentage of Fat-free Mass) | Pre and Post 12-week Intervention
  Fat-free mass (percentage of total body weight, %) was estimated using multifrequency bioelectrical impedance with an 8-electrode device (TANITA-MC780MA, Tanita Corp., Tokyo, Japan) after at least 8 hours of fasting. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants wore light clothing and were asked to urinate immediately before the measurement.
Assessed changes in Anthropometry: Perimeters | Pre and Post 12-week Intervention
  Waist circumference (cm) was measured at the midpoint between the lower lateral margin of the 10th rib and the iliac crest, perpendicular to the longitudinal axis of the trunk. Abdominal circumference (cm) was measured at the level of the umbilicus, perpendicular to the longitudinal axis of the trunk. Hip circumference (cm) was measured at the level of the greatest posterior prominence of the buttocks, perpendicular to the longitudinal axis of the trunk. Thigh circumference (cm) was measured at the midpoint between the greater trochanter and the lateral tibial condyle. All measurements were performed with the participant standing upright, and relaxed. Each measurement was taken twice, and a third measurement was performed if the difference exceeded 1%. The mean of the two most similar records was registered.
Assessed changes in Anthropometry: Waist to Hip Ratio | Pre and Post 12-week Intervention
  Waist-to-hip ratio (WHR) was calculated as waist circumference (cm) divided by hip circumference (cm).
Assessed changes in Anthropometry: Skinfold thickness | Pre and Post 12-week Intervention
  Thigh skinfold thickness was measured at two-thirds of the distance from the iliospinale point (the lowest part of the anterior superior iliac spine) to the superolateral border of the patella, over the belly of the vastus lateralis muscle. Measurements were taken on the dominant leg. Two measurements were obtained, and a third was taken if the difference between the first two exceeded 5%. The mean of the two most similar records was recorded.

SECONDARY OUTCOMES:
Assessed changes in dietary intake: Frequency of consumption | Pre and post the 12-week intervention
  One week before laboratory measurements, participants completed a 7-day weighed food record, including two weekend days, to capture habitual dietary intake. Additionally, dietary habits were assessed through a 137-item semi-quantitative Food Frequency Questionnaire (FFQ), previously validated in a Mediterranean Spanish population. The FFQ was administered in face-to-face interviews by trained nutritionists and included information on vitamin/mineral supplements and alcohol consumption. Participants reported their habitual intake over the previous year using a 9-level frequency scale (ranging from "never or almost never" to ">6 times/day").
Assessed changes in dietary intakes: 24 hours dietary recalls | Pre and post the 12-week intervention
  Nutrient intakes were estimated using the DIAL software for Windows (version 1.19; Ortega et al., 1999), a validated tool for quantitative and qualitative assessment of dietary intake in the Spanish population. The software converted food consumption into daily energy and nutrient values, expressed absolute intake (g/day), percentage of Recommended Intake (RI) coverage, and the energy distribution profile (percentage of total energy from proteins, fats, carbohydrates, and alcohol).
Assessed changes in dietary intakes: Mediterranean Diet Adherence | Pre and post the 12-week intervention
  Adherence to the Mediterranean Diet was evaluated using a validated 14-item questionnaire for the Spanish population (3), with scores ranging from 0 (lowest adherence) to 14 (highest adherence). The resulting score was classified into three categories: low adherence (range: 0-5), moderate adherence (range: 6-9), and high adherence to MedDiet (range: 10-14).
Assessed changes in accelerometry: Physical activity time | Pre and post the 12-week intervention
  Physical activity and inactivity will be assessed using triaxial accelerometers (GENEActiv; ActivInsights Ltd., Kimbolton, UK) placed on the non-dominant wrist for at least six consecutive days (direct method). Participants will be instructed to wear the device at all times, including during sleep and water-based activities, to ensure comprehensive data capture. Valid data will be defined as a minimum wear of 16 hours per day for at least four days (three weekdays and one weekend day) following established protocols (10.1177/07334648231218095). Accelerometers will be set to 60 Hz (10.1111/sms.12795, 10.1249/MSS.0000000000000289). Raw data will be downloaded using GENEActiv software version 3.3 and processed using the GGIR package (version 3.0.9) in R (v4.1.1, R Core Team, Vienna, Austria), which auto-calibrates the data based on local gravity and calculates the Euclidean Norm Minus One (ENMO) to minimize sensor calibration error (https://doi.org/10.1152/japplphysiol.00421.2014).
Assessed changes in physical activity and sedentary time | Pre and post the 12-week intervention
  Physical activity, sedentary time, and sleep will also be estimated through self-reported questionnaires, using the International Physical Activity Questionnaire Short Version (IPAQ-SF), previously validated in Spain. The IPAQ-SF will provide estimates of sedentary time, moderate and vigorous activity in minutes per week.
Assessed changes in Resting Energy Expenditure | Pre and post the 12-week intervention
  After at least 8 hours of fasting, resting energy expenditure was estimated by indirect calorimetry. Participants were instructed the day before testing to maintain their usual lifestyle, refrain from alcohol or caffeine for 24 hours, and avoid vigorous physical activity for 72 hours. Participants lay supine for 30 minutes wearing a mask connected to a gas analyzer (open circuit, Jaeger MasterScreen CPX® (CareFusion, San Diego, USA)). The resting rates of fat and carbohydrate oxidation were used to determine the resting energy expenditure in kcal per minute (kcal/min).
Assessed changes in Maximal Fat Oxidation | Pre and post the 12-week intervention
  Maximal fat oxidation was determined through a gradual test on a cycloergometer (Lode Excalibur, Groningen, Netherlands). Gas exchange (VO2, VCO2, RER) was recorded using indirect calorimetry (Jaeger MasterScreen CPX®), and heart rate was measured continuously over the test with Polar Team 2 (Polar Electro Inc., Lake Success, NY). The test consisted of a starting load of 15W with increments of 15W every 3 minutes until the respiratory quotient reached a stable value of 1. Throughout the test, a cadence of 60 r.p.m. was maintained. Fat oxidation (g/min) values were estimated from oxygen and carbohydrate data averaged over the last minute of each 3-minute stage, using the Frayn stoichiometric equation, and then the higher fat oxidation value was recorded.
Assessed changes in Relative Intensity of Maximal fat Oxidation during exercise | Pre and post the 12-week intervention
  The relative intensity of maximal fat oxidation (FatMax) reflects the exercise intensity (% of maximal oxygen consumption (VO2max)) at which fat oxidation reaches its peak. FatMax was determined from the graded maximal fat oxidation (MFO) cycling test in a cyclo-ergometer (Lode Excalibur, Groningen, Netherlands). The test started at 15 W with 15-W increments every 3 min until the respiratory quotient reached 1, maintaining 60 rpm. Gas exchange (VO2, VCO2, RER) was measured via indirect calorimetry (Jaeger MasterScreen CPX®), and heart rate was continuously monitored (Polar Team 2, Polar Electro, NY). After the MFO test, a second incremental test with 15W/min increments until exhaustion from the last load of MFO test was performed to determine VO2max. Fat oxidation rates (g/min) were calculated using the Frayn equation and plotted against relative VO2 (%VO2max). The VO2 corresponding to maximal fat oxidation was identified as FatMax.
Assessed changes in Cardiorespiratory Fitness | Pre and post the 12-week intervention
  Maximal oxygen consumption (VO2max, ml/min) was assessed using an incremental test on a cycle ergometer (Lode Excalibur) following the maximal fat oxidation (MFO) test. Gas exchange (VO2, VCO2, and RER) was recorded using an indirect calorimeter (Jaeger MasterScreen CPX®), and heart rate was measured continuously over the test with Polar Team 2 (Polar Electro Inc). After a 5-min rest following the MFO test, the VO2max phase started at the last workload achieved in the MFO stage and increased by 15 W every minute, maintaining a pedaling cadence of 70-90 rpm until volitional exhaustion. Maximal effort was confirmed when at least three of the following criteria were met: a VO2 plateau (VO2-time slope <0.05 L·min-1 during the last 30 s), ≥90% of age-predicted maximal heart rate, a respiratory exchange ratio (RER) ≥1.10, perceived exertion of 8-10 on the Borg scale, and volitional fatigue. If fewer than three criteria were reached, the VO2 value was recorded as VO2peak.
Assessed changes in self-reported quality of life | Pre and post the 12-week intervention
  Self-reported quality of life will be registered by applying the Short Form 36-health survey (SF-36) questionnaire previously validated in Spain. The SF-36 is a generic measure of quality of life and has been evaluated for a wide variety of medical conditions, including diabetes. The SF-36 includes 36 questions that evaluate 8 subscales, scores for each scale range from 0 to 100, with higher scores indicating higher level of function or wellbeing. The physical component summary is derived from the 4 subscales of physical functioning, role physical, bodily pain, and general health; while the mental component summary is derived from the subscales of vitality, social functioning, role emotional, and mental health.
Assessed changes in blood pressure | Pre and post the 12-week intervention
  Systolic and diastolic blood pressures will be recorded three times by using the validated Omron HEM 742 blood pressure monitoring device with the participant seated, back supported in chair and feet flat on floor without legs crossed, after they rested 5 minutes. The guidelines of the Hypertension and Cardiology European Societies and the Spanish one will be used to classify blood pressure stages of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Casals, PhD, Principal Investigator — University of Cadiz; Jesús Ponce González, PhD, Principal Investigator — University of Cadiz
Locations (1):
- Science of Education Faculty, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No